CLINICAL TRIAL: NCT06977230
Title: The Effect of Remote Ischemic Preconditioning on Myocardial Protection in Patients With Type 2 Diabetes Mellitus Undergoing Coronary Artery Bypass Graft Surgery: A Randomized Controlled Double-Blind Study
Brief Title: Remote Ischemic Preconditioning in Type 2 Diabetic Patients Undergoing CABG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Melike Korkmaz Toker, Associate Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RIPC-T2DM-CABG-2025
Record Dates: First submitted 2025-05-07; First posted 2025-05-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus; Coronary Artery Bypass; Remote Ischaemic Conditioning
Keywords: High sensitive Troponin T; Diabetes mellitus Type 2; Coronary Artery Bypass; Myocardial Ischemia; Remote Ischemic Conditioning; Acute Kidney Injury; Cardioprotection
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Myocardial Ischemia; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Preconditioning Group (Active Comparator): Patients randomized to this group will receive remote ischemic preconditioning (RIPC) prior to sternotomy. RIPC will be performed by inflating a blood pressure cuff on the upper limb to 200 mmHg for 5 minutes, followed by 5 minutes of deflation. This cycle will be repeated 5 times before the start of cardiopulmonary bypass.Assigned Intervention: Remote Ischemic Preconditioning
  Interventions: Procedure: Remote Ischemic Preconditioning
- Control Group (No Intervention): Patients in the control group will undergo standard anesthetic and surgical care without the application of remote ischemic preconditioning.

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — Remote ischemic preconditioning (RIPC) will be performed after anesthesia induction and before surgical incision. A standard blood pressure cuff will be placed on the upper limb (without arterial cannulation), inflated to 200 mmHg for 5 minutes, and then deflated for 5 minutes. This cycle will be repeated five times prior to sternotomy. The procedure will be carried out under general anesthesia, ensuring patient blinding. No pharmacological agents are involved in this intervention
  Arms: Remote Ischemic Preconditioning Group

SUMMARY:
This randomized, double-blind, prospective clinical trial aims to investigate the effect of remote ischemic preconditioning (RIPC) on myocardial protection in patients with type 2 diabetes mellitus undergoing elective coronary artery bypass graft (CABG) surgery. Perioperative myocardial injury remains a significant concern during CABG, particularly in high-risk patients such as those with diabetes. RIPC is a low-cost, non-invasive intervention that may reduce myocardial damage by enhancing ischemic tolerance through intermittent limb ischemia.

Sixty patients aged 40-85 years with type 2 diabetes scheduled for isolated CABG will be randomized to either receive RIPC or standard care. RIPC will be applied through five cycles of upper limb cuff inflation and deflation prior to sternotomy. High-sensitivity troponin T levels will be measured at 24, 48, and 72 hours postoperatively to assess myocardial injury. Secondary outcomes include acute kidney injury (KDIGO classification), maximum vasoactive-inotropic score (VIS) during the first 72 postoperative hours, ICU and hospital length of stay. This study will provide insight into the cardioprotective role of RIPC in diabetic patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus and receiving medical treatment
* Scheduled for isolated elective coronary artery bypass graft (CABG) surgery
* American Society of Anesthesiologists (ASA) physical status class III or IV
* Age between 40 and 85 years

Exclusion Criteria:

Emergency CABG surgery Reoperation (revision surgery) Left ventricular ejection fraction (LVEF) < 40% History of cardiac arrest or cardiogenic shock Pregnancy Clinically significant peripheral arterial disease affecting the upper limbs Hepatic dysfunction (bilirubin > 20 μmol/L or INR > 2.0) Renal failure (eGFR < 20 mL/min/1.73 m²) Ongoing treatment with glibenclamide or nicorandil (agents known to interfere with ischemic preconditioning mechanisms) Asthma

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative 24-hour high-sensitivity Troponin T level | 24 hours after surgery
  Myocardial injury will be assessed by measuring high-sensitivity cardiac Troponin T (hs-TnT) levels at 24 hours after coronary artery bypass graft (CABG) surgery. Blood samples will be collected at the 24th postoperative hour and analyzed using a standardized high-sensitivity Troponin T assay (reference range: 0-14 ng/L). The primary endpoint will be the mean hs-TnT concentration in each group.

SECONDARY OUTCOMES:
Incidence and severity of acute kidney injury | Within 72 hours postoperatively
Postoperative 48-hour high-sensitivity Troponin T level | 48 hours after surgery
  Myocardial injury will be assessed by measuring high-sensitivity cardiac Troponin T (hs-TnT) levels at 48 hours after coronary artery bypass graft (CABG) surgery. Blood samples will be collected at the 48th postoperative hour and analyzed using a standardized high-sensitivity Troponin T assay (reference range: 0-14 ng/L). The primary endpoint will be the mean hs-TnT concentration in each group.
Postoperative 72-hour high-sensitivity Troponin T level | 72 hours after surgery
  Myocardial injury will be assessed by measuring high-sensitivity cardiac Troponin T (hs-TnT) levels at 72 hours after coronary artery bypass graft (CABG) surgery. Blood samples will be collected at the 72th postoperative hour and analyzed using a standardized high-sensitivity Troponin T assay (reference range: 0-14 ng/L). The primary endpoint will be the mean hs-TnT concentration in each group.
Maximum vasoactive-inotropic score (VIS) in the first 72 hours postoperatively | 0-72 hours after surgery
Length of ICU and hospital stay | From ICU admission to ICU discharge and from hospital admission to hospital discharge, assessed up to 60 days

OTHER OUTCOMES:
Correlation between high-sensitivity Troponin T levels and maximum vasoactive-inotropic score (VIS) | Within 72 hours after surgery
Correlation between Troponin T levels and duration of ICU stay | From ICU admission through ICU discharge
Correlation between intraoperative maximum vasoactive-inotropic score (VIS) and postoperative myocardial injury | Intraoperative period and up to 72 hours postoperatively
  The correlation between the maximum intraoperative VIS score and high-sensitivity Troponin T (hs-TnT) levels measured at 24, 48, and 72 hours postoperatively will be assessed. This outcome will evaluate whether intraoperative hemodynamic support requirement is associated with subsequent myocardial injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) may not be shared due to institutional policies and ethical considerations regarding patient confidentiality. The study protocol does not include provisions for public data sharing, and participants dmay not provide consent for external access to their personal health data.